CLINICAL TRIAL: NCT04047992
Title: "The Effects of Exoskeletal-Assisted Walking on Seated Balance Using the Indego™"
Brief Title: Seated Balance Using the Indego™
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ann M. Spungen, EdD, Associate Director, VA RR&D National Center for the Medical Consequences of Spinal Cord Injury, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPU-17-029
Record Dates: First submitted 2018-05-15; First posted 2019-08-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Exoskeleton Users (Experimental): All participants will receive 36 sessions of supervised EAW training using Indego™ for 12 weeks (3 to 4 sessions per week, 4-6 hours per week). The goal is to complete all 36 sessions in 12 weeks, but allowing for a two-week carryover to accommodate schedule conflicts or missed sessions.
  Interventions: Device: Indego™ Exoskeleton

INTERVENTIONS:
Device: Indego™ Exoskeleton — The Indego® is a powered exoskeleton that can be used as a mode of therapy in an institutional setting. Proper walking in this device requires the user to manipulate their center of gravity and balance by postural trunk excursions in order for the legs to take steps.

SUMMARY:
Exoskeleton-assisted walking (EAW) provides a new mobility option and appears to have potential therapeutic benefits for persons with SCI. However, present day technology is not sufficient to replace the wheelchair. During EAW, users stand upright, maintain static and dynamic balance by actively and passively stimulating trunk and lower limb muscles in a manner not challenged during wheelchair use. Preliminary results in our laboratory suggest that the indirect balance challenges and postural perturbations that result during EAW training transfer to better seated balance control, resulting in more independence during seated activities. The purpose of this pilot study is to determine the effects of EAW training on various measures of seated balance (primary outcomes) and body composition (secondary outcomes). Twenty people with SCI (T4 and below) who are wheelchair users for mobility and cannot walk independently will be recruited. The participants will receive 36 sessions of EAW training in 12 weeks. The outcomes will be evaluated pre (baseline) and post (24 and 36 sessions). If EAW devices can be demonstrated to help people with SCI have better seated balance, in addition to the other potential benefits that are being investigated elsewhere, then exoskeletons may have the possibility to be more readily accepted in the clinical, home environments, and by the insurance companies.

DETAILED DESCRIPTION:
Introduction/Background: People with spinal cord injury (SCI) can lose partial to complete voluntary control of arm, trunk and leg muscles, resulting in an inability to sit with stability, stand and/or walk. Because of poor trunk control during sitting, it may be challenging to reach for objects, dress or transfer independently, and the risk of a fall from their wheelchair is increased. Exoskeleton-assisted walking (EAW) provides upright, over ground mobility and has been demonstrated to be beneficial to improve patient-reported quality of life and some health-related outcomes. However, present day exoskeletons are not ready to replace the wheelchair. Our preliminary findings suggest that while walking in an exoskeleton, people with SCI are challenged to maintain upright balance by using their trunk muscles in a way that is rarely done from a wheelchair. Stimulation of the trunk muscles from upright postural challenges during EAW appears to benefit overall seated trunk control.

Summary of Goals and Objectives: The purpose of this study is to determine whether EAW can improve the primary outcomes of: seated balance, seated activities of daily living, and trunk muscle use. Additional secondary outcomes for body composition will be studied. Twenty people with SCI (T4 and below) who are wheelchair users will be recruited to participate.

Impact: The investigators believe that EAW training will significantly improve seated balance to improve wheelchair safety, stability and quality of life, thus, empowering people with SCI who use a wheelchair to live more independently. If EAW is demonstrated to have a significant benefit on seated balance, then use of these devices in the clinical and home environments may be further justified.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic or non-traumatic SCI ≥6 months duration of SCI;
2. Wheelchair-user for indoor and outdoor mobility;
3. Level and completeness of injury T4 and below with complete or incomplete SCI (ISNCSCI A to D);
4. Able to hold the crutches in hands with or without modifications; and
5. Able to provide informed consent.

Exclusion Criteria:

1. Diagnosis of neurological injury other than SCI;
2. Progressive condition that would be expected to result in changing neurological status;
3. Severe concurrent medical disease, illness or condition judged to be contraindicated by the Site Physician;
4. Anthropocentric incompatibility to be fitted with the device;
5. Traumatic or high impact lower extremity fracture within the past 2 years;
6. Fragility, minimal trauma or low impact fracture of the lower extremity since spinal cord injury;
7. Knee BMD < 0.60 gm/cm2;
8. Total hip BMD T-scores < -3.5;
9. Untreatable severe spasticity judged to be contraindicated by the Site Physician;
10. Flexion contracture that is incompatible with the device;
11. Limitations in ankle range of motion that cannot be adapted with an orthotic device (plantar flexion > 00);
12. Fracture of the foot by x-ray and confirmed by CT;
13. Untreated or uncontrolled hypertension (systolic blood pressure >140 mmHg; diastolic blood pressure >90 mmHg);
14. Unresolved orthostatic hypotension (systolic blood pressure <90 mmHg; diastolic blood pressure <60 mmHg) as judged to be contraindicated by the Site Physician;
15. Current pressure ulcer of the arms, trunk, pelvic area, or lower extremities;
16. History of seizure;
17. Use of medications that significantly lower seizure threshold, such as tricyclic antidepressants, amphetamines, neuroleptics, dalfampridine, and bupropion;
18. History of stroke, brain tumor, brain abscess, or multiple sclerosis;
19. History of moderate or severe head trauma (loss of consciousness for greater than one hour or evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging);
20. History of implanted brain/spine/nerve simulators, aneurysm clips, ferromagnetic metallic implants, or cardiac pacemaker/defibrillator;
21. Psychopathology documentation in the medical record or history that may conflict with study objectives; and/or
22. Pregnancy or women who plan to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Seated Computerized Dynamic Posturography (sCDP) | Change from baseline after 8 weeks and after 12 weeks.
  Seated balance will be measured by assessment of the limits of stability (LOS) using computerized dynamic posturography (SMART EquiTest, Natus). The SMART EquiTest® system utilizes a dynamic force plate to quantify the vertical forces exerted through the participant's center of gravity as s/he sits on a cushioned block with back unsupported and arms crossed over the clavicles.

SECONDARY OUTCOMES:
Seated Activities of Daily Living (ADLs) | Change from baseline after 8 weeks and after 12 weeks.
  Participants' seated ADLs will be assessed by self-reported Spinal Cord Independence Measure (SCIM) and Spinal Cord Injury - Functional Index (SCI-FI, short forms). Participants' functional performance of ADLs will be assessed using the timed t-shirt dressing test by a study team member.
Motor Evoked Potentials (MEPs) | Change from baseline after 8 weeks and after 12 weeks.
  Leg muscles will be used to assess neuroplastic changes between the motor cortex and descending neural pathways below incomplete spinal lesions.

OTHER OUTCOMES:
Spinal Cord Independence Measure (SCIM) | Change from baseline after 8 weeks and after 12 weeks.
  The SCIM is a clinical tool to evaluate the independent performance of ADL especially for people with SCI.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided